CLINICAL TRIAL: NCT04028154
Title: Comparison of Erector Spinae Plane (ESP) Block and Thoracolumbar Interfascial Plane(TLIP) Block for the Management of Postoperative Pain in Spinal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, SINEM SARI, M.D., clinical research, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020/06
Record Dates: First submitted 2019-07-16; First posted 2019-07-22 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Parapsychology; Dental Occlusion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESP Block (Experimental)
  Interventions: Procedure: Erector Spinae Plane (ESP) Block
- TLIP Block (Active Comparator)
  Interventions: Procedure: Thoracolumbar interfacial plane (TLIP) Block

INTERVENTIONS:
Procedure: Erector Spinae Plane (ESP) Block — ESP Block: Bilateral ESP block and with ultrasound guidance will be applied A total 40 ml, 20 ml bupivacaine 0.5%, 20 ml saline.
  Arms: ESP Block
Procedure: Thoracolumbar interfacial plane (TLIP) Block — TLIP Block: BilateralTLIP block and with ultrasound guidance will be applied A total 40 ml, 20 ml bupivacaine 0.5%, 20 ml saline.
  Arms: TLIP Block

SUMMARY:
Lumbar vertebra surgery is one of the most common surgical procedures. After lumbar veretebra surgery, patients complain of excessive pain. Postoperative pain usually occurs in the early postoperative period and delays patient mobilization and thus lengthens hospital stay.

The aim of this study was to compare the efficacy of erector spina plan(ESP) block and thoraco lumbar interfacial(TLIP) block on postoperative pain in patients with spinal surgery.

DETAILED DESCRIPTION:
Plan blocks are used as a good and safe option for multimodal analgesia techniques in postoperative pain control in spinal surgery.

The ESP block was first described in 2016 for the treatment of thoracic neuropathic pain.

In the following process; ESP block has been reported to provide effective postoperative analgesia in thoracic and breast surgery, bariatric surgery and upper abdominal surgery.

Finally, ESP block has been reported to provide effective postoperative analgesia in veretebra surgeries.

The mechanism of ESP analgesic action has been demonstrated in cadaver studies where injected local anesthetics are caused by diffusion of the spinal nerves into the ventral and dorsal ramycin by spreading in the cranial and caudal directions.

ESP block relieves incisional pain by creating an effective block in a wide area of the posterior, lateral and anterior thoracic and lumbar walls.

In addition, ESP block prevents visceral autonomic pain and provides good postoperative analgesia.

The thoracolumbar interfacial plan block (TLIP) is the other para-spinal plan block.

In this ultrasound guided block, local anesthetic targets the dorsal branches of the thoracolumbar nerves by spreading between the facies of the multifidus and longissimus muscles at the 3rd lumbar spine.

In this way, it has been reported to provide effective analgesia in spinal surgeries.

Routine ultrasonography guided ESP block or TLIP blog was planned randomly. Peroperative analgesia plan will be applied to all patients in the same way. In this protocol intravenous paracetamol was 1 g and tramadol was 1 mg / kg. Paracetamol and tramadol infusions are then administered every eight hours.

Postoperative analgesia protocol: At the end of the operation, pain levels will be recorded by the Numeric Rating Scale (NRS) system at 30 minutes, 1.6, 12, and 24 hours after the first admission to the recovery room.

Tramadol PCA and paracetamol were administered to the patient every eight hours.

During the follow-up of the patient, it is planned to continue NRS follow-up. In this period, intramuscular 75 mg diclofenac sodium will be administered if NRS is 4 or above.The amount of analgesia consumption, recovery analgesia needs and times will be noted in detail.

When the patient is mobilized and discharged will be recorded.

The aim of this study was to compare the efficacy of erector spina plan(ESP) block and thoraco lumbar interfacial(TLIP) block on postoperative pain in patients with spinal surgery.

ELIGIBILITY:
Inclusion Criteria:

* 68 patients
* ASA I-III,
* Aged 18-75 years
* underwent lumbar spine surgery under elective conditions

Exclusion Criteria:

* Presence of contraindications to LA agents used in this study
* Use of chronic opioids,
* Psychiatric disorders.
* The presence of infection at the injection area.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
NRS(numerical rating scala) | [Time Frame: 24 hours]
  Each item is scored 0-10 ( 0=no pain, 10= pain as bad as can be) Postoperative pain intensity reported with NRS score : 30. minute, 1. hours, 6. hours, 12. hours, 24. hours
pruritus | [Time Frame: 24 hours]
  each criterion is reported as present or absent each criterion is reported as present or absent
mobilized | [Time Frame: 7 days]
  each criterion is reported as when the patient is mobilized
nausea and vomiting | [Time Frame: 24 hours]
  each criterion is reported as present or absent each criterion is reported as present or absent
use of antiemetics | [Time Frame: 24 hours]
  each criterion is reported as present or absent each criterion is reported as present or absent
discharged | [Time Frame: 7 days]
  each criterion is reported as when the patient is discharged

CONTACTS AND LOCATIONS:
Overall Officials: Sinem Sarı, Principal Investigator — Aydin Adnan Menderes University
Locations (1):
- Adnan Menderes University Medical Faculty, Anesthesiology and Reanimation Department, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Almeida CR, Oliveira AR, Cunha P. Continuous Bilateral Erector of Spine Plane Block at T8 for Extensive Lumbar Spine Fusion Surgery: Case Report. Pain Pract. 2019 Jun;19(5):536-540. doi: 10.1111/papr.12774. Epub 2019 Mar 15. PMID 30758122